CLINICAL TRIAL: NCT00157690
Title: A Multicentre, Double-Blind, Randomized Placebo-Controlled Study of 70mg Alendronate Once Weekly for the Prevention and Treatment of Osteoporosis in Canadian Adult Cystic Fibrosis Patients
Brief Title: Study of Alendronate to Prevent and Treat Osteoporosis in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); London Health Sciences Centre (Other); University of Calgary (Other); McGill University (Other); Laval University (Other); Merck Frosst Canada Ltd. (Industry)
Responsible Party: Dr. Alexandra Papaioannou, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MK-0217 Protocol 214
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Cystic Fibrosis; Osteoporosis; Bone Diseases, Metabolic
Keywords: Alendronate; Bisphosphonates; Cystic Fibrosis; Osteoporosis
MeSH Terms: conditions — Cystic Fibrosis; Osteoporosis; Bone Diseases, Metabolic | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Alendronate
  Interventions: Drug: Alendronate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alendronate — 70 mg 1x weekly for 12 months
  Other Names: Fosamax
  Arms: 1
Drug: Placebo — 70 mg 1 x weekly for 12 months
  Arms: 2

SUMMARY:
The primary objective of this study is to determine efficacy of 70 mg alendronate once weekly compared to placebo. This will be measured by percent changes in lumbar spine(LS) bone mineral density(BMD) in adult cystic fibrosis(CF)patients after one year of treatment. The investigators hypothesize that in adult CF patients with osteopenia or osteoporosis, alendronate 70 mg once weekly will produce a mean increase from baseline in lumbar spine BMD that is greater than that observed with placebo at 12 months.

DETAILED DESCRIPTION:
Randomized controled trial have begun to establish the efficacy and safety of bisphosphonates in CF patients with decreased BMD. The development of a once weekly dosing regimen of alendronate and the low prevalence of esophageal adverse events may be an advantageous therapeutic option for this high-risk population. This is a one-year randomized, double-blind, placebo-controlled, multicentre study in 55 CF patients with osteopenia or osteoporosis. Six Canadian centres are participating in this study. Patients randomized to treatment will receive 70 mg oral alendronate once weekly, while controls will receive identical placebo once weekly. All medication dispensed will be concealed. There will be no dose modification during the course of the trial. All patients will receive a total of 1000 mg calcium, 500 through supplementation and 500 through diet. All patients will continue to take vitamin D supplementation ( 2 tablets per day, 400 IU vitamin D/tablet).

ELIGIBILITY:
Inclusion Criteria:

1. CF; confirmed by a positive sweat test or DNA analysis
2. age 18 years or above at the time of informed consent
3. osteopenia (-2.5< BMD t-score<1.0) or osteoporosis (BMD t-score <-2.5)t-score at the LS (1-4)or total hip
4. provision of informed consent

Exclusion Criteria:

1. endoscopy-proven esophagitis, gastritis, ulceration, or abnormalities of the esophagus which delay esophageal emptying such as stricture, achalasia, or esophageal varices
2. significantly impaired renal function; this is defined as serum creatinine >177 umol/L
3. current or recent (within 1 year prior to randomization) consumption of an excess of alcohol or abuse of drugs; an excess of alcohol is defined as more than four of any of the following per day, or a combination of more that four of the following per day: 30 mL distilled spirits, 240 mL beer, or 120 mL wine
4. history of prior organ transplantation
5. any condition which may interfere with the evaluation of LS BMD as determined in a screening radiograph by a radiologist at the central facility e.g. spinal fusion, confluent aortic calcifications, surgical artefact, excessive osteophytes, or other permanent artefact; hip prostheses or any other condition that may interfere with the evaluation of hip BMD
6. participation in another clinical trial 30 days prior to enrolment or within 6 half-lives of the study drug if applicable
7. pregnancy, lactation, or a desire to become pregnant; safe effective birthcontrol must be used
8. know hypersensitivity or abnormal reaction to study drug or other bisphosphonates
9. use of drugs know to affect bone within 6 months of starting trial medication (e.g. thiazide, diuretics, calcitonin, calcitriol, anabolic steroids, estrogen or estrogen-related drugs (e.g. tamoxifen, raloxifene, tibolone high dose vaginal estrogen), progesterone, fluoride: this does not include the birth control pill
10. patients currently receiving another bisphosphonate in whom treatment efficacy has been established; only patients who are intolerant to or did not respond to another bisphosphonate will be considered for inclusion; patients must have ceased treatment with any bisphosphonate for at least 1 year prior to enrolment
11. use of systemic corticosteroids at a dose of at least 7.5 mg/day or greater within last 6 months
12. concomitant use of any investigational drug other than the study medication
13. current or recent (within 1 year prior to randomization) metabolic bone disorders other than secondary osteoporosis, such as Paget's disease, renal osteodystrophy, osteomalacia (25-OHD<25nmol/L), hypoparathyroidism, hyperparathyroidism; TSH outside normal laboratory range, with values that are assessed as clinically significant by the investigator; if on replacement therapy, dose should be stable and TSH within normal range for a minimum of 6 weeks prior to trial enrolment
14. hypocalcemia from any cause, corrected for low albumin
15. any history of cancer; for relatively benign skin malignancies, such as basal cell carcinoma or squamous cell carcinoma and patients with a history of successfully treated cervical carcinoma in istu, a documented six-month remission is required before study entry
16. poor medical or psychiatric risk for treatment with an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-12; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine efficacy of 70 mg alendronate once weekly compared to placebo, measured by changes in LS BMD in adult CF patients after one year of treatment | 12 months

SECONDARY OUTCOMES:
To determine the efficacy of 70 mg alendronate once weekly compared to placebo measured by percent changes in total hip BMD, proximal femur BMD, and N-telopeptide at one year in adult CF patients. | 12 months
To determine health-related quality of life (HRQL) using the SF-36 instrument. | 12 months
To determine HRQL using the Cystic Fibrosis Questionnaire (CFQ). | 12 months
To determine the safety of 70 mg of alendronate given once weekly compared with placebo in adult CF patients | 12 months
To determine correlations between BMD and patient characteristics, including but not limited to the following: corticosteroid use, height, weight, body mass index BMI) and forced expired volume in 1 minute (FEV1). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, M.D., Principal Investigator — McMaster University; Andreas Freitag, M.D., Study Chair — McMaster University; Jonathan D Adachi, M.D., Study Chair — McMaster University
Locations (6):
- Canada (6):
  - Dr. Harvey Rabin - Health Sciences Centre, Calgary, Alberta
  - McMaster University, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Centre de Recherche - CHUM, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - CHUL Hospital, Sainte-Foy, Quebec

REFERENCES:
- [Background] Aris RM, Lester GE, Caminiti M, Blackwood AD, Hensler M, Lark RK, Hecker TM, Renner JB, Guillen U, Brown SA, Neuringer IP, Chalermskulrat W, Ontjes DA. Efficacy of alendronate in adults with cystic fibrosis with low bone density. Am J Respir Crit Care Med. 2004 Jan 1;169(1):77-82. doi: 10.1164/rccm.200307-1049OC. Epub 2003 Oct 16. PMID 14563654
- [Background] Aris RM, Merkel PA, Bachrach LK, Borowitz DS, Boyle MP, Elkin SL, Guise TA, Hardin DS, Haworth CS, Holick MF, Joseph PM, O'Brien K, Tullis E, Watts NB, White TB. Guide to bone health and disease in cystic fibrosis. J Clin Endocrinol Metab. 2005 Mar;90(3):1888-96. doi: 10.1210/jc.2004-1629. Epub 2004 Dec 21. PMID 15613415
- [Derived] Papaioannou A, Kennedy CC, Freitag A, Ioannidis G, O'Neill J, Webber C, Pui M, Berthiaume Y, Rabin HR, Paterson N, Jeanneret A, Matouk E, Villeneuve J, Nixon M, Adachi JD. Alendronate once weekly for the prevention and treatment of bone loss in Canadian adult cystic fibrosis patients (CFOS trial). Chest. 2008 Oct;134(4):794-800. doi: 10.1378/chest.08-0608. Epub 2008 Jul 18. PMID 18641106